CLINICAL TRIAL: NCT01491412
Title: RECONNECT-S GAMMA : A Non-interventional Study to Observe Real-life Usage of Atypical Antipsychotics in the Acute Inpatient Management of Schizophrenia
Brief Title: Non-interventional Study: Real-life Use of Atypical Antipsychotics in Acute Inpatient Management of Schizophrenia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NME-SER-2011/1
Record Dates: First submitted 2011-12-09; First posted 2011-12-14 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Acute Psychotic Episode; Schizophrenia
Keywords: Schizophrenia; antipsychotics; real life treatment; non-interventional
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute psychotic episode in schizophrenia: Subjects suffering from schizophrenia being discharged from the hospital following hospitalisation due to acute psychotic episode

SUMMARY:
This is an observational study describing the real-life antipsychotic treatment during the hospitalisation of the patients due to acute psychotic episode.

In this NIS subject's data will be collected at one visit at the moment of discharge from the hospital.

The results of the study would help to characterise the discrepancy between current clinical practice and treatment guidelines, indicating that atypical antipsychotics are preferable and should be used in monotherapy during acute psychotic episodes in subjects with schizophrenia. Available evidence have revealed a frequent use of first-generation antipsychotics, polypharmacy, intramuscular route of administration and use of atypical antipsychotics in doses lower than recommended in registered summary of product characteristics.

DETAILED DESCRIPTION:
RECONNECT-S GAMMA : A non-interventional study to observe real-life usage of atypical antipsychotics in the acute inpatient management of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent has been obtained from the Subject and/or his/her legal representative (as per local regulatory requirements).
* Meet the diagnostic criteria for schizophrenia stated in The Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria
* Subject is hospitalised due to an acute psychotic episode

Exclusion Criteria:

* Current participation in any clinical trial.
* Previous enrolment in the present NIS (in case of recurrence occurred during the enrolment period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from schizophrenia being discharged from the hospital following hospitalisation due to acute psychotic episode
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2011-12; Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Description of used atypical antipsychotic(s) during hospitalisation | hospitalisation period, an expected average of 2 weeks (variable per patient)
  The data will be collected at one visit at the moment of discharge from the hospital.
Description of the daily dosage of atypical antipsychotic(s) during hospitalisation | hospitalisation period, an expected average of 2 weeks (variable per patient)
  The data will be collected at one visit at the moment of discharge from the hospital.
Description of mode of administration of atypical antipsychotic(s) during hospitalisation | hospitalisation period, an expected average of 2 weeks (variable per patient)
  The data will be collected at one visit at the moment of discharge from the hospital.

SECONDARY OUTCOMES:
Percent of patients with atypical antipsychotic as monotherapy | hospitalisation period, an expected average of 2 weeks (variable per patient)
Percent of patients with combinations of antipsychotics. | hospitalisation period, an expected average of 2 weeks (variable per patient)
Description of main criteria used for selection of an antipsychotic during hospitalisation. | hospitalisation period, an expected average of 2 weeks (variable per patient)
Description of the usage of psychometric scales in day to day practice, to evaluate the disease symptoms and thus the efficacy of treatment. | hospitalisation period, an expected average of 2 weeks (variable per patient)
Description of used concomitant psychiatric medication (other than atypical antipsychotic) during the hospitalization | hospitalisation period, an expected average of 2 weeks (variable per patient)
Description of the relationship between medication used during the hospitalization and maintenance therapy recommended upon discharge | hospitalisation period, an expected average of 2 weeks (variable per patient)
Description of the study population by collecting the following exploratory variables: demographic, educational, economical, social data, psychiatric and somatic health. | hospitalisation period, an expected average of 2 weeks (variable per patient)

CONTACTS AND LOCATIONS:
Overall Officials: Radu TEODORESCU, Prof., Principal Investigator — Spitalul Clinic of Psychiatry named after Prof. Dr. Alexandru Obregia, Romania
Locations (14):
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kistarcsa
  - Research Site, Nyíregyháza
  - Research Site, Szekszárd
  - Research Site, Székesfehérvár
- Latvia (5):
  - Research Site, Daugavpils
  - Research Site, Jelgava
  - Research Site, Liepāja
  - Research Site, Riga
  - Research Site, Strenči
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Iași